CLINICAL TRIAL: NCT03250663
Title: Eucrisa for Atopic Dermatitis: Measuring and Improving Adherence to Topical Eucrisa in Patients With Atopic Dermatitis
Brief Title: Eucrisa for Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00045841
Record Dates: First submitted 2017-08-04; First posted 2017-08-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Mild to Moderate Atopic Dermatitis
Keywords: topical therapy, atopic dermatitis,
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Intervention Model Description: All subjects will receive study medication. Groups will be randomized to receive online treatment response surveys.
Who Masked: Participant, Investigator
Masking Description: adherence data of the randomized subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Standard of Care (Active Comparator): Subjects receive study medication, EUCRISA (crisaborole) ointment 2%, and follow standard of care
  Interventions: Drug: EUCRISA
- Arm 2 - Online Treatment Response (Experimental): Subjects receive study medication, EUCRISA (crisaborole) ointment 2%, and electronic treatment response emails
  Interventions: Behavioral: Online Treatment response; Drug: EUCRISA

INTERVENTIONS:
Behavioral: Online Treatment response — Electronic treatment response survey to track use of study medication, EUCRISA (crisaborole) ointment 2%.
  Arms: Arm 2 - Online Treatment Response
Drug: EUCRISA — Participants are given EUCRISA (crisaborole) ointment 2%.

SUMMARY:
Patients with mild to moderate atopic dermatitis will be asked to participate in helping the study team determine how well the medication works for atopic dermatitis. Participants will not be told that adherence will be monitored. Patients will be dispensed topical crisaborole 2% ointment (Eucrisa®) in a medication tube fitted with a Medication Event Monitoring System (MEMS) cap if they agree to participate. This cap records dates and times the bottle is opened and this data can be downloaded and tabulated with the associated software.

Investigators and subjects will be blinded to the adherence data until the final treatment (12 month) session. The study subjects will be randomized to two groups. After baseline visit, both groups will come for a follow-up visit at 1 month, 3 months, 6 months, and 12 months. The intervention group will also be asked to complete an online treatment response survey designed to improve adherence at weekly intervals for 6 weeks, then monthly thereafter.

The study will consist of a 12-month Treatment Phase. Study subjects will be instructed to apply the medication twice daily (morning and evening) to all of their AD lesions. They will be instructed to apply the smallest amount of study medication possible that is sufficient to cover all lesions. These instructions are standard-of-care for patients with AD.

Subjects will be asked to bring their medication tubes with them at each visit. At each visit, the study coordinator will weigh the medication tube and download the MEMS cap data. Disclosure of the adherence monitoring will occur at the 12 month visit (or end of treatment), at which time the results of the subject's adherence behavior will be used to supply individualized treatment options for each subject (feedback session).

At each visit, drug tubes will be measured for weight to determine the amount of study medication used. This data will be correlated with the extent of BSA involved and the response of the disease. The MEMS caps will be downloaded at each visit.

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) affects between 10% and 30% of all children, making it one of the most common childhood diseases. Recent epidemiological studies report a trend toward the increasing prevalence of AD in children. Symptoms of AD include dry, scaly, and intensely itchy skin. A number of treatments are available for these patients. Topical corticosteroids are commonly prescribed. Topical immunomodulators without the potential for steroid atrophy are also used. A non-steroidal topical, Eucrisa (crisaborole) ointment, is specifically indicated for mild to moderate atopic dermatitis and was approved for marketing in the U.S. for the treatment atopic dermatitis in December 2016. The 2% ointment is approved for use in patients ages 2 and older. Unfortunately, many people with atopic dermatitis do not adequately respond to topical treatment.

It is widely recognized that adherence to oral medications is poor. Adherence to medication in chronic disease is worse. Adherence to topical medication for chronic disease in children is horrible. In a previous study, the investigator found that the adherence of children to topical triamcinolone for atopic dermatitis was poor. Adherence dropped by roughly 60-70% over the first 3 days of treatment. While that study analyzed adherence over 8 weeks, the long-term adherence to topical treatment in patients with atopic dermatitis is not well characterized.

Measures to improve adherence have the potential to improve treatment outcomes. Adherence to topical treatment tends to improve around the time of office visits (so called, "white coat compliance"), much as tooth flossing behavior improves around the time of dental visits. Standard-of-care treatment of atopic dermatitis generally involves having patients return in roughly 4 weeks to assess treatment efficacy. Clinical trials generally have more frequent visits. The investigator's recent studies have suggested that adherence may be improved with virtual medical visits, alleviating the need for more frequent in-person office visits that can be costly and negatively impact access to care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 2-64.
* Stable or worsening atopic dermatitis affecting 5% or greater body surface area. Face and genital areas can be included in the body surface area determination and treatment area.
* The ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
* The ability to understand and sign a written informed consent/assent form, which must be obtained prior to treatment.

Exclusion Criteria:

* Known allergy to crisaborole or to any component of the formulations.
* The use of systemic therapy for atopic dermatitis within the past 4 weeks.
* Use of prescription topical therapy for atopic dermatitis (e.g., corticosteroids or retinoids) within the past 2 weeks.
* Use of any investigational therapy within the past 4 weeks.
* Pregnant females, females who are breast feeding, or females of childbearing potential who are not practicing an acceptable method of birth control (abstinence, birth control pill/patch, barrier with spermicidal jelly, IUD, etc.), as determined by the investigator. Acceptable contraception must be used during the entire study. A pregnancy test will be performed on females of childbearing potential at baseline and at 6 month and 12 month.
* Any other condition, which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.

Ages: 2 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Adherence to topical Therapy | 12 months
  Difference in adherence between standard-of-care and intervention with use of the impact of an internet reporting intervention on adherence. Asking 50% of the enrolled subjects to complete internet-based surveys on their use of the study medication.

SECONDARY OUTCOMES:
Adherence to topical therapy #1 | 12 months
  Difference in adherence between standard-of-care and intervention with use of MEMS Caps: The Medical Events Monitoring System (MEMS) by MWV formerly Aardex Corporation in Switzerland will be used. The MEMS incorporates a microprocessor into the cap of a standard medication tube. Each time the tube is opened for at least 3 seconds, the time and date are recorded. The Eucrisa 2% ointment will be fitted with a MEMS cap using a specially designed adaptor. Subjects will be asked to bring the unused portion of the medication tube to each visit so that the medication can be "checked and redispensed". At each visit the information is downloaded via the MEMS communicator onto a computer database by the study staff to ensure the blinding of the primary physician performing the severity measures.
Adherence to topical therapy #2 | 12 months
  Difference in adherence between standard-of-care and intervention with use of Eczema Area and Severity Index (EASI): Disease severity will be assessed by a physician with the Eczema Area and Severity Index (EASI). This measure is a commonly used and well-validated instrument of eczema severity. It is weighted for area in each of the four body regions (which differs for adults and children under 7) and scores erythema, excoriation, induration/papulation, and lichenification. The total scores range from 0-72.
Adherence to topical therapy #3 | 12 months
  Difference in adherence between standard-of-care and intervention with use Visual Analog Scale (VAS) for Itching. A 100mm VAS will be used to measure itch intensity at each visit. VAS is a self-report tool that is designed to present to the respondent a rating scale with minimum constraints. VAS data is recorded as the number of mm from the left of the line with the range 0-100mm. The Visual Analog Scale is anchored with the verbal descriptions of "no itching" on the left and "the most intense itching imaginable" on the right. VAS is considered a useful tool for the measurement of symptoms such as itch.
Adherence to topical therapy #4 | 12 months
  difference in adherence between the standard-of-care and intervention with use of the Investigator Global Assessment(IGA) This measure is commonly used as a quick and simple way to quantify disease severity both for clinical studies and in a non-study clinic setting. Score ranges from '0' = clear or "No inflammatory signs of AD" to '4' = Very Severe Disease with "severe erythema and severe papulation/infiltration with oozing/crusting

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay C Strowd, MD, FAAD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Heath Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Study team does not plan to make individual participant data available; only the total outcome

DOCUMENTS (1):
  • Informed Consent Form (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT03250663/ICF_000.pdf